CLINICAL TRIAL: NCT07092436
Title: Pediatric Upper-Limb Rehabilitation With PhiCube, a Modular Bilateral End-Effector Device.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto di Sistemi e Tecnologie Industriali Intelligenti per il Manifatturiero Avanzato (Other)
Collaborators: IRCCS Fondazione Stella Maris (Other); IRCCS Eugenio Medea (Other); Fondazione Don Carlo Gnocchi Onlus (Other); IRCCS Fondazione Istituto Neurologico Mondino Pavia (Unknown); Ospedale IRCCS G. Gaslini di Genova (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PhiCube-Pediatric
Record Dates: First submitted 2025-07-02; First posted 2025-07-29 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Congenital and Acquired Neuromotor Disorders; Developmental Coordination Disorder (DCD)
Keywords: Pediatric Rehabilitation; Upper Limb Rehabilitation; Robotic Rehabilitation; Bilateral Training; Neuromotor Disorders
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PhiCube Bilateral Upper Limb Rehabilitation (Experimental)
  Interventions: Device: Robotic bilateral upper limb rehabilitation training

INTERVENTIONS:
Device: Robotic bilateral upper limb rehabilitation training — Bilateral upper limb rehabilitation using PhiCube, a modular robotic end-effector device with two motorized axes that can assist or resist patient movements. Treatment consists of 30 sessions over 3 months (3 sessions/week, 45 minutes each) combining motor training with gaming elements specifically designed for pediatric populations. The device's modular design allows customization for individual patient needs and bilateral coordination training. Sessions focus on improving range of motion, precision, dexterity, and movement fluidity through controlled, repetitive, high-intensity exercises in children aged 4-18 years with neuromotor disorders and developmental coordination disorder.

SUMMARY:
The present investigation is configured as a multicenter clinical study in a within-group pilot phase.

This study aims to investigate primarily the feasibility of use and effectiveness of a treatment for upper limb function in children aged 4 to 18 years with congenital and acquired neuromotor disorders through a new portable robotic system, called PhiCube, designed for bilateral neuromotor rehabilitation of the upper limbs in subjects with neuromotor disorders.

In order to specifically investigate also the potential impact of PhiCube on movement planning aspects, the study will also involve a small group of children aged 4 to 18 years with Developmental Coordination Disorder (DCD).

Before (PreT0 and T0) and after (T1 and T2) treatment, standardized assessment tests will be administered. Regarding the investigation objectives reported above, the primary outcome measure will be the Melbourne Assessment-2 (MA2), a standardized, valid and reliable instrument for evaluating the quality of upper limb movement in children with neurological deficits, capable of measuring four elements of movement quality: range of motion, accuracy, dexterity and fluency. As secondary outcome measures, Abilhand-Kids has been chosen, a brief questionnaire that measures 21 main daily bimanual activities completed by the parent or caregiver, and various subtests and questionnaires aimed at evaluating the neuropsychological processes involved and the effects related to auditory feedback perception.

The treatment will have a total duration of approximately 3 months and will be organized in 3 weekly sessions lasting 45 minutes each, to reach a total of 30.

Descriptive statistics of the clinical and technological variables obtained in the evaluation and rehabilitation phases will be calculated. Subsequently, treatment efficacy analyses through the robotic device are planned, comparing pre-post clinical variables. All collected data will finally be analyzed in order to compare the rehabilitative efficacy of the device with respect to the different groups of participants identified based on diagnostic profile.

ELIGIBILITY:
Inclusion Criteria:

* For subjects with congenital and acquired neuromotor disorders:

  * Diagnosis of congenital and acquired neuromotor disorders
  * Age between 4 and 18 years at the time of recruitment
  * Modified Ashworth Scale (MAS) less than 3
  * MACS level I-IV
  * Sufficient capacity to understand the proposed activities
  * Availability to attend the facility
* For subjects with developmental coordination disorder (DCD):

  * Diagnosis of developmental coordination disorder (DCD)
  * Age between 4 and 18 years at the time of recruitment
  * Sufficient capacity to understand the proposed activities
  * Availability to attend the facility

Exclusion Criteria:

* For subjects with congenital and acquired neuromotor disorders:

  * Severe sensory deficits
  * Onset of pathologies that prevent participation
  * Worsening of pre-existing comorbidities
* For subjects with developmental coordination disorder (DCD):

  * Severe sensory deficits
  * Onset of pathologies that prevent participation
  * Worsening of pre-existing comorbidities

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Upper limb movement quality in children with neurological deficits | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  Quality of upper limb movement in children with neurological deficits, measured through Melbourne Assessment-2 (MA2), which is able to measure four elements of movement quality: range of motion, precision, dexterity and fluidity.

SECONDARY OUTCOMES:
ABILHAND-Kids Questionnaire | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  A brief questionnaire measuring 21 main bimanual daily activities. Scores are assigned by parents based on the child's difficulty in performing daily activities, with a 3-point scale (impossible, difficult, easy).
Leiter-3 Sustained Attention Subtest | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  A subtest of the Leiter-3 non-verbal cognitive scale that evaluates sustained visual attention through tasks of increasing complexity within a specific time period. The number of correctly selected target elements is recorded.
NEPSY-II Inhibition Subtest | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  Evaluates inhibitory control abilities of automatic verbal responses through administration of 3 different conditions for two different stimulus sets, requiring naming, inhibition with reversal, and alternating responses based on color.
NEPSY-II Auditory Attention Subtest | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  Assesses the ability to maintain sustained attention to auditory stimuli performance and inhibit automatic motor responses in two tasks of increasing complexity with incremental executive control demands.
NEPSY-II Manual Posture Imitation subtest | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  This subtest assesses the child's ability to accurately imitate a series of progressively complex hand and finger postures demonstrated by the examiner. The raw score is obtained by summing the number of correctly executed postures, separately recorded for the dominant and non-dominant hands. From the total raw score, a weighted score is derived, which in turn is used to calculate the standard score based on normative data.
NEPSY-II Manual Motor Sequences subtest | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  This subtest evaluates the child's ability to observe and reproduce sequences of hand movements demonstrated by the examiner. The sequences become progressively more complex and require the integration of motor planning, attention, and imitation abilities. The raw score is calculated by summing the number of correctly imitated sequences. From the total raw score, a weighted score is derived, which is then converted into a standard score based on normative data.
NEPSY-II Arrow subtest | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  This subtests evaluates the ability to judge line orientation considering direction, distance, orientation, and angularity. The task requires the integration of visual attention, orientation discrimination, and mental rotation.
  The raw score is obtained by summing the number of correct responses across all items. From this total raw score, a weighted score is calculated and then converted into a standard score based on age-specific normative data.
NEPSY-II Route Finding subtest | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  This subtest assesses the ability to use a small schematic map to locate targets on a larger schematic map.
  The raw score corresponds to the number of correctly identified routes. From this raw score, a weighted score is derived and then transformed into a standard score using normative tables based on the child's age.
BRIEF P/2 Questionnaire | Assessed at 4 time points: - PreT0: 2 months before treatment initiation - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period - T2: 1 month after treatment completion
  Parent-administered questionnaire evaluating executive functions in daily life contexts. Parents rate behaviors on a 3-point Likert scale based on frequency over the past six months.
Usability questionnaire | T1: Immediately after completing the treatment period
  Custom questionnaire administered to stakeholders (children and operators) at treatment completion to investigate system usability.
Acceptability questionnaire | T1: Immediately after completing the treatment period
  Custom questionnaire administered to stakeholders (children and operators) at treatment completion to investigate system acceptability.
Compliance questionnaire | T1: Immediately after completing the treatment period
  Custom questionnaire administered to stakeholders (children and operators) at treatment completion to investigate child and operator compliance.
Movement smoothness | - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period
  Measures of how continuous and even a movement is, without sudden stops or changes in speed. It is measured by the normalized jerk.
Trajectory error | - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period
  Measures the error made by one limb in following a proposed trajectory via the screen.
Bilateral coordination | - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period
  Measures coordination between limbs in performing the same movement simultaneously by calculating the difference between axes coordinates.
Audio Feedback Effect Evaluation | - T0: Immediately before starting PhiCube treatment - T1: Immediately after completing the treatment period
  Assessment of how audio feedback influences motivational and satisfaction aspects through three interaction conditions (no feedback, reward feedback, help feedback) using VAS scales for fun and engagement, adapted In-game Questionnaire, and open-ended questions about the child's experience.